CLINICAL TRIAL: NCT01616888
Title: Rug Eluting Balloon With Paclitaxel for Treatment of In-stent Restenosis in Femoropopliteal Arteries
Brief Title: Paclitaxel Eluting Balloon for SFA In-stent Restenosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KTT2
Record Dates: First submitted 2012-06-07; First posted 2012-06-12 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: In-stent Arterial Restenosis
Keywords: drug eluting balloon with paclitaxel; in stent restenosis; femoropopliteal arteries; angioplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment arm (Active Comparator): SFA angioplasty with In.Pact Admiral drug eluting balloon
  Interventions: Device: PTA with drug eluting balloon with paclitaxel

INTERVENTIONS:
Device: PTA with drug eluting balloon with paclitaxel — Angioplasty with drug eluting balloon with paclitaxel on femoropopliteal arteries
  Other Names: In.Pact Admiral by Medtronic

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy on the use of drug eluting balloon (DEB) with paclitaxel to treat in-stent restenosis in femoropopliteal arteries.

DETAILED DESCRIPTION:
Peripheral artery disease (PAD) in the lower extremities can cause claudication, pain in the legs or feet and slowly wounds that can affect patients' quality of life and increase the risk of leg amputation and death. Both conventional balloon angioplasty (CBA) alone and CBA plus bare metal stents are the current primary endovascular therapy to treat PAD. However, exaggerated neointimal hyperplasia leading to in-stent restenosis is associated with CBA. Paclitaxel coated balloons have been recognized to be safe and effective for the treatment of coronary in-stent restenosis, which the investigators hypothesize to be applicable in femoropopliteal cases.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* chronic symptomatic lower limb ischemia defined as Rutherford categories 2, 3, 4 or 5
* in-stent restenosis or occlusion in SFA or PPA 20mm - 200mm

Exclusion Criteria:

* participation in another investigational drug or device trial
* life expectancy less than 12 months
* acute ischemia and/or acute thrombosis of the SFA/PPA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-06; Primary Completion 2015-06 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Target lesion patency at 6-month follow-up. | 6-month post index procedure
  Patency of target lesion at 6-month follow-up based on duplex ultrasound.

SECONDARY OUTCOMES:
Clinical success up to 12 months post index procedure | 12 months post index procedure
  Improvement on clinical evaluations including staging of PAD according to the Rutherford category, ABI at 1, 6, 12 months post procedure compared to baseline assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Kong Teng Tan, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada